CLINICAL TRIAL: NCT05326152
Title: Intralesional or Intramuscular Hepatitis B Vaccine Versus Intralesional Saline in the Treatment of Multiple Common Warts
Brief Title: Intralesional Versus Intramuscular Hepatitis B Vaccine Immunotherapy for Warts
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Basma Magdy Elkholy, MD, Clinical professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB# 6547/-25-11-2020
Record Dates: First submitted 2022-02-15; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Intralesional Versus Intramuscular Hepatitis B Vaccine for Multiple Common Warts
MeSH Terms: interventions — GeneVac B

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IntralesionaL Hepatitis B vaccine (Experimental): 0.2 ml of hepatitis B vaccine injected in the largest wart and repeated every 2 weeks till clearance of warts or for a maximum of 5 sessions
  Interventions: Biological: hepatitis B vaccine immunotherapy of common warts (GeneVac-B 10 ml vial, Serum Institute of India Ltd., Pune, India)
- Intramuscular Hepatitis B vaccine (Experimental): 0.5 ml injected in the deltoid muscle for those who were younger than 19 years at the time of study and 1 ml for those who were 20 years and older at the time of study.
  Three injections were done at 0, 1, and 4 months.
  Interventions: Biological: hepatitis B vaccine immunotherapy of common warts (GeneVac-B 10 ml vial, Serum Institute of India Ltd., Pune, India)
- Intralesional saline (Placebo Comparator): 0.2 ml of saline injected in the largest wart and repeated every 2 weeks till clearance of warts or for a maximum of 5 sessions
  Interventions: Biological: Intralesional saline

INTERVENTIONS:
Biological: hepatitis B vaccine immunotherapy of common warts (GeneVac-B 10 ml vial, Serum Institute of India Ltd., Pune, India) — Randomized placebo-controlled comparative effectiveness clinical trial
  Arms: IntralesionaL Hepatitis B vaccine; Intramuscular Hepatitis B vaccine
Biological: Intralesional saline — Intralesional saline
  Arms: Intralesional saline

SUMMARY:
Assessment of the effectiveness of intralesional and intramuscular hepatitis B vaccine in treatment of multiple common warts.

DETAILED DESCRIPTION:
Recently, intralesional immunotherapy by different antigens, including Candida antigen and purified protein derivative PPD has been proved effective in the treatment of different types of warts. Hepatitis B vaccine is one of the DNA vaccines that are regarded as being potentially safer, relatively cheap and easy to produce with no special storage requirements because they are extremely stable and allow for potential simultaneous immunization against multiple antigens or pathogens via co-expression of multiple epitopes on single plasmid. Hepatitis B vaccine could be a promising immunotherapeutic vaccine in the field of intralesional immunotherapy of warts. Moreover, the efficacy of intramuscular injection of hepatitis B vaccine would be assessed and compared to its intralesional injection.

ELIGIBILITY:
Inclusion Criteria:

• Adult patients of both sexes with multiple (> 3 warts) common warts of various sites, sizes and duration, with or without distant warts after taking informed consent from all patients

Exclusion Criteria:

* Pregnancy or lactation.
* Serious systemic or anaphylactic reaction to a prior dose of the vaccine or to any of its components.
* Allergic skin disorders such as generalized eczema and urticaria.
* Moderate or severe acute illness with or without fever.
* Previous wart therapy within 1 month prior to the study.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Efficacy of intralesional versus intramuscular hepatitis B vaccine in the treatment of multiple common warts | up to 3 months after last injection
  Percentage of patients showing complete response to intralesional hepatitis B vaccine and intramuscular hepatitis B vaccine.
  Complete response: complete disappearance of warts including distant warts and complete return of normal skin markings (100%).
  Partial response: if the warts have regressed in size by 50-99%. No response: less than 50% decrease in wart size.
Immediate adverse effects | up to 20 minutes after intralesional or intramuscular injection of vaccine

SECONDARY OUTCOMES:
Efficacy of intralesional versus intramuscular hepatitis B vaccine in distant wart response | up to 3 months
  Percentage of patients showing complete response of their distant warts to intralesional hepatitis B vaccine and intramuscular hepatitis B vaccine.
  Complete response: complete disappearance of distant warts and complete return of normal skin markings (100%).
  Partial response: if the distant warts have regressed in size by 50-99%. No response: less than 50% decrease in distant wart size.
Late adverse effects | up to 6 months follow-up period
Recurrence | for 6 months-follow-up
  after complete clearance of all warts

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided